CLINICAL TRIAL: NCT04970147
Title: Development of Evidence-Based Nursing Care Bundle in Gastrostomy Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Rana Elcin SEZER CEREN, Principal Investigator, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KA-21029
Record Dates: First submitted 2021-07-16; First posted 2021-07-21 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Nervous System Diseases
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- there are not arm for this study. (Other): there is not a control group for this study.
  Interventions: Other: Gastrostomy care bundle

INTERVENTIONS:
Other: Gastrostomy care bundle — Gastrostomy care bundle

SUMMARY:
The concept of care bundle; It was developed by the American Institute for Healthcare Improvement (IHI) in 2001 to provide the best care safely in order to achieve desired results in patient care, increase compliance with standard procedures, improve patient safety and quality of care. Ensuring that nurses perform gastrostomy care correctly and according to the guidelines published in international standards will minimize the development of problems that may arise in gastrostomy care. The aim of this study was to development and implementation the gastrostomy care bundle for gastrostomy care.

DETAILED DESCRIPTION:
The concept of care bundle; It was developed by the American Institute for Healthcare Improvement (IHI) in 2001 to provide the best care safely in order to achieve desired results in patient care, increase compliance with standard procedures, improve patient safety and quality of care. Ensuring that nurses perform gastrostomy care correctly and according to the guidelines published in international standards will minimize the development of problems that may arise in gastrostomy care.

Method: The research was planned as a mixed type research design in order to development and implementation the gastrostomy care bundle for gastrostomy care. The study was planned to be carried out in Hacettepe University Adult Hospital Brain and neurosurgery intensive care unit between September 2021 and September 2022. In the quantitative phase of the research; The development of the gastrostomy care bundle will be carried out using the care bundle development approach in line with the recommendations of the Institute for Healthcare Improvement (IHI) and expert opinions will be taken. Nurses working in the brain and neurosurgery intensive care unit will be trained on the gastrostomy care bundle and will be expected to practice care bundle. Before the training, nurses will be asked to fill in the "Nurse Introductory Information Form", "Evidence-Based Attitude Scale towards Nursing" and "Gastrostomy Care Questionnaire (pre-test)". The nurse population of the research will consist of 14 nurses working in the brain and neurosurgery intensive care unit. At this stage, the sample selection will not be made, and it will be tried to reach all of the working nurses. The "Gastrostomy Care bundle" form will be used by the nurses in the gastrostomy care in the brain and Neurosurgery intensive care unit between September 2021 and September 2022 , which is determined for the patient sample. Nurses' compliance with the care bundle will be evaluated by the researcher with the "Gastrostomy Care Bundle Compliance Evaluation Control Form" by making daily visits to the intensive care unit. At the end of the period determined for the use of the care bundle in the intensive care unit, the nurses will be asked to fill in the "Evidence-Based Attitude Scale towards Nursing" and "Gastrostomy Care Questionnaire (post-test)". In the qualitative phase of the research, nurses working in the brain and neurosurgery intensive care unit will be interviewed about their experiences with the use of gastrostomy care bundle. At the end of the study, nurses' compliance with the use of care bundle, the effect of gastrostomy care bundle use/gastrostomy education on nurses' knowledge levels and attitudes towards evidence-based nursing, and nurses' views on gastrostomy care bundle will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

For the patient;

* Patients with gastrostomy over the age of 18 who receive treatment and care in the brain and neurosurgery intensive care unit, For the nurse;
* Nurses working in the brain and neurosurgery intensive care unit,

Exclusion Criteria:

* For the patient;
* Patients who are treated in the brain and neurosurgery intensive care unit but do not have gastrostomy,
* Patients under the age of 18,
* Not giving consent to the study. For the nurse;
* Leaving the brain and neurosurgery intensive care unit before the work process is completed,
* Not filling out data collection forms at any stage of the study,
* Not participating in the semi-structured in-depth individual interview,
* Not giving consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Compliance with the use of the care bundle | 6 months
  Nurses' compliance with the use of the care bundle will be considered successful if the rate in the calculation is 95% or more
Knowledge levels of nurses about gastrostomy care | 6 months
  Data to be obtained from the Gastrostomy Care Questionnaire (pre-test) to be administered before the training to be given to nurses for the evidence-based nursing, gastrostomy, gastrostomy care bundle, and the Gastrostomy Care Questionnaire (post-test) to be administered after the training and use of the gastrostomy care bundle.
Attitude Scale towards Evidence-Based Nursing | 6 months
  Data to be obtained from the "Attitude Scale towards Evidence-Based Nursing" to be administered before the training to be given to the nurses for the evidence-based nursing, gastrostomy and gastrostomy care bundle, and the "Attitude Scale towards Evidence-Based Nursing" to be administered after the training and the use of the gastrostomy care bundle a survey using a 5-point Likert scale.

SECONDARY OUTCOMES:
Nurses' views on the use of care bundle | 6 months
  "For the Use of Gastrostomy Care Bundle" to be conducted with nurses in order to evaluate the post-application views of the nurses who applied the care bundle.

CONTACTS AND LOCATIONS:
Overall Officials: Rana Elcin SEZER CEREN, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided